CLINICAL TRIAL: NCT06470139
Title: Pericapsular Nerve Group (PENG) Block with Ropivacaine Vs Ropivacaine and Dexamethasone in Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: Dexamethasone for PENG Block in Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6/2024
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy; Hip Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine (Active Comparator): Ultrasound-guided PENG block - 20ml 0,2% ropivacaine + 2ml 0.9% NaCl
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Ropivacaine+Dexamethasone (Active Comparator): Ultrasound-guided PENG block - 20ml 0,2% ropivacaine + 4mg Dexamethasone
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution + 4mg Dexamethasone

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — 20ml 0.2% Ropivacaine + 2.0ml 0.9% NaCl
  Arms: Ropivacaine
Drug: Ropivacaine 0.2% Injectable Solution + 4mg Dexamethasone — 20ml 0.2% Ropivacaine + 4mg Dexamethasone
  Arms: Ropivacaine+Dexamethasone

SUMMARY:
Effect of adding Dexamethasone to Periarticular Nerve Group Block in Patients undergoing Total Hip Arthroplasty

DETAILED DESCRIPTION:
Hip arthroplasty is one of the most common orthopaedic procedures, especially in elderly patients, due to the deformation of joints. Patients may complain of severe pain due to surgical trauma and prostheses. Regional anaesthesia methods may be performed to reduce the inflammatory response, opioid consumption, and opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total hip arthroplasty
* patients aged >65 and <100 years
* patients able to provide informed consent
* patients able to reliably report symptoms to the research team

Exclusion Criteria:

* inability to provide first-party consent due to cognitive impairment or a language barrier

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Total Opioid Consumption | 48 hours after surgery
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 4 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 8 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 12 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 24 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 48 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating
Nerve damage | 12 hours after surgery
  Nerve damage assesent will be performed using scale: N0- no nerve damage; N1- minor - sensory paresthesia; N2- majorcomplete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome
Nerve damage | 24 hours after surgery
  Nerve damage assesent will be performed using scale: N0- no nerve damage; N1- minor - sensory paresthesia; N2- majorcomplete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome
Nerve damage | 48 hours after surgery
  Nerve damage assesent will be performed using scale: N0- no nerve damage; N1- minor - sensory paresthesia; N2- majorcomplete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome
glucose | 24 hours after surgery
  blood glucose levels
glucose | 12 hours after surgery
  blood glucose levels
glucose | 48 hours after surgery
  blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Domagalska, M.D. Ph.D., Study Chair — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: Yes